CLINICAL TRIAL: NCT05096065
Title: An Open-label Dose-finding Study to Evaluate the Pharmacodynamic (PD) Profiles and Efficacy of Different Dosing Regimens of Leuprolide Oral Tablets (Ovarest®) in Women With Endometriosis
Brief Title: Study to Evaluate the Pharmacodynamics and Efficacy of Leuprolide Tablets (Ovarest®) in Women With Endometriosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Enteris BioPharma Inc. (Industry)
Collaborators: Parexel (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LOPDT-ENDO-02
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Endometriosis
Keywords: Leuprolide oral tablets; Endometriosis; pharmacodynamic
MeSH Terms: conditions — Endometriosis | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A: Leuprolide Oral Tablet, 120 mg QD (Experimental): Leuprolide Oral Tablet (Ovarest), 120 mg (2 x 60 mg tablets), administered once daily (QD), for up to 35 consecutive days with food-intake restrictions.
  Interventions: Drug: Leuprolide Oral Tablet - 120 mg - QD- Treatment A
- Treatment B: Leuprolide Oral Tablet, 80 mg QD (Experimental): Leuprolide Oral Tablet (Ovarest), 80 mg (2 x 40 mg tablets), administered once daily (QD) for up to 35 consecutive days with food-intake restrictions.
  Interventions: Drug: Leuprolide Oral Tablet - 80 mg - QD - Treatment B
- Treatment C: Leuprolide Oral Tablet, 60 mg QD (Experimental): Leuprolide Oral Tablet (Ovarest), 60 mg, administered once daily (QD) for up to 29 consecutive days with food-intake restrictions.
  Interventions: Drug: Leuprolide Oral Tablet - 60 mg - QD - Treatment C
- Treatment D: Leuprolide Oral Tablet, 60 mg BID (Experimental): Leuprolide Oral Tablet (Ovarest), 60 mg, administered twice daily (BID), 12 hours apart for up to 35 consecutive days with food-intake restrictions.
  Interventions: Drug: Leuprolide Oral Tablet - 60 mg - BID - Treatment D
- Treatment E:Leuprolide Oral Tablet (Ovarest), 40 mg BID (Experimental): Leuprolide Oral Tablet (Ovarest), 40 mg, administered twice daily (BID), 12 hours apart for up to 29 consecutive days with food-intake restrictions.
  Interventions: Drug: Leuprolide Oral Tablet - 40 mg - BID - Treatment E

INTERVENTIONS:
Drug: Leuprolide Oral Tablet - 120 mg - QD- Treatment A — If the subject during Treatment "A" meets the pharmacodynamic success criterion (estradiol level <20 pg/mL on Treatment Day 29 of the First Treatment Cycle), in the Second Treatment Cycle, she will be assigned Treatment "B" - 80 mg (2 x 40 mg tablets) (QD), with food-intake restrictions.
  If the subject during Treatment "A" fails to meet the pharmacodynamic success criterion (i.e., if estradiol level ≥20 pg/mL on Treatment Day 29 of the First Treatment Cycle), then she will be switched to the Second Treatment Cycle with Treatment "D" - 60 mg (BID) with food intake restrictions.
  Other Names: Ovarest® 60 mg
  Arms: Treatment A: Leuprolide Oral Tablet, 120 mg QD
Drug: Leuprolide Oral Tablet - 80 mg - QD - Treatment B — If the subject on Treatment "B" meets the pharmacodynamic success criterion (estradiol level <20 pg/mL on Treatment Day 29 of the Second Treatment Cycle), then she will be switched to the Third Treatment Cycle with Treatment "C" - 60 mg (QD) with food-intake restrictions.
  If the subject on Treatment "B" does not meet the pharmacodynamic success criterion (i.e., if estradiol level ≥20 pg/mL on Treatment Day 29 of the Second Treatment Cycle), then she will be switched to the Third Treatment Cycle with Treatment "E" - 40 mg (BID) with food intake restrictions.
  Other Names: Ovarest® 40 mg
  Arms: Treatment B: Leuprolide Oral Tablet, 80 mg QD
Drug: Leuprolide Oral Tablet - 60 mg - QD - Treatment C — For up to 29 consecutive days with food-intake restrictions
  Other Names: Ovarest® 60 mg
  Arms: Treatment C: Leuprolide Oral Tablet, 60 mg QD
Drug: Leuprolide Oral Tablet - 60 mg - BID - Treatment D — If the subject on Treatment "D" fails to meet the pharmacodynamic success criterion (i.e., if estradiol level ≥20 pg/mL on Treatment Day 29 of the Second Treatment Cycle), she will be discontinued from the study following completion of the Second Treatment Cycle.
  If the subject during Treatment "D" meets the pharmacodynamic success criterion (estradiol level <20 pg/mL on Treatment Day 29 of her Second Treatment Cycle), then she will be switched to the Third Treatment Cycle with Treatment "E" - 40 mg (BID) with food intake restrictions.
  Other Names: Ovarest® 60 mg
  Arms: Treatment D: Leuprolide Oral Tablet, 60 mg BID
Drug: Leuprolide Oral Tablet - 40 mg - BID - Treatment E — For up to 29 consecutive days with food-intake restrictions
  Other Names: Ovarest® 40 mg
  Arms: Treatment E:Leuprolide Oral Tablet (Ovarest), 40 mg BID

SUMMARY:
The pharmacodynamic endpoint of percentage of subjects with suppressed estradiol level (less than 20 pg/mL) on cycle day 29 is the primary endpoint of the study.

DETAILED DESCRIPTION:
Objectives of this study:

1. To determine efficacy and pharmacodynamic effects of various dosing regimens of Ovarest® (within the 60-mg - 120 mg daily dosing range) in women with endometriosis.
2. To determine a minimally effective daily dosing regimen of Ovarest® with pharmacodynamic effects at least comparable to the historical data for marketed Lupron Depot formulations and for GnRH antagonists indicated for the treatment of endometriosis.
3. To evaluate safety and tolerability of the long-term administration of leuprolide within the targeted daily dosing range in women with endometriosis.

The most important goal of this study is to provide adequate dose-response data for the suppression of estradiol (E2) levels below the menopausal threshold of 20 pg/mL. Results of this study in conjunction of Enteris proprietary PK data will support further development of Leuprolide Acetate Oral Tablet for the treatment of reproductive disorders, particularly endometriosis. Another reason for this trial is to support a comparative evaluation of the PD effects across the QD and BID regimens delivering the same overall dose of Ovarest

ELIGIBILITY:
Inclusion criteria:

1. Women diagnosed with endometriosis and having pelvic pain, both treatment naive or previously treated with GnRH agonists or antagonists with improvement
2. Premenopausal females in general good health, including absence of current COVID infection (positive test or presence of symptoms), aged 18 to 49 years
3. BMI ≥18 and ≤35 kg/m2, and weight ≥110 lb. (≈50 kg).
4. A documented estradiol level ≥ 40 pg/mL at screening or on retest
5. Regular menstrual cycles with a usual length ranging from 21 days to 35 days. If subject has recently used hormonal birth control, historical data prior to use will be used to determine qualification and must also meet this criterion.
6. If of childbearing potential and sexually active with a risk of pregnancy, willing to use acceptable methods of contraception (Note: acceptable methods of contraception are specified in Section 8.1)
7. Willing to refrain from excessive use of alcohol during the entire study and willing to refrain from use of alcohol 24 hours prior to any PK blood draw taken during the study
8. Willing to refrain from the use of any hormone-containing or hormone-altering substances during the study.
9. Willing and able to adhere to medication schedule and to utilize the AiCure medication adherence monitoring platform correctly with the administration of each dose of medication throughout the duration of the 3 treatment cycles comprising this study
10. Willing and capable to give informed consent to participate in study

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

1. Hypersensitivity to GnRH, GnRH agonist analogs, similar nonapeptides, or any of the excipients in LUPRON DEPOT. Note: This is a contraindication from the Lupron Depot label.
2. Undiagnosed abnormal vaginal bleeding. Note: This is a contraindication from the Lupron Depot label.
3. Known or suspected pregnancy, or subjects who are considering becoming pregnant prior to the conclusion of this study. Note: LUPRON DEPOT is contraindicated in women who are or may become pregnant while receiving the drug. LUPRON DEPOT may cause fetal harm when administered to a pregnant woman…. If this drug is used during pregnancy, or if the patient becomes pregnant while taking this drug, the patient should be apprised of the potential hazard to the fetus.
4. Breastfeeding or within 2 months after stopping breastfeeding (relative to the screening visit). Note: Use of LUPRON DEPOT is contraindicated in women who are breastfeeding.
5. Thrombophlebitis, thromboembolic disorders, cerebral apoplexy, or a past history of these conditions. Note: Per the LUPRON DEPOT label, a possible coadministration of norethindrone acetate is contraindicated in women with thrombophlebitis, thromboembolic disorders, cerebral apoplexy, or a past history of these conditions.
6. Markedly impaired liver function or liver disease. Note: Per the LUPRON DEPOT label, a possible coadministration of norethindrone acetate is contraindicated in women with markedly impaired liver function or liver disease.
7. Known or suspected carcinoma of the breast. Note: Per the LUPRON DEPOT label, a possible coadministration of norethindrone acetate is contraindicated in women with known or suspected carcinoma of the breast.
8. Status postpartum or postabortion within a period of 2 months prior to the screening visit
9. History of significant alcohol or drug abuse within one year prior to the screening visit
10. Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mm Hg, diastolic blood pressure lower than 50 or over 90 mm Hg, or heart rate less than 50 or over 100 bpm) at screening (following recheck after five minutes at rest)
11. Any clinically significant history or presence of neurologic, endocrinologic, pulmonary, hematologic, immunologic, or metabolic disease
12. History of severe respiratory depression or pulmonary insufficiency
13. Diabetes mellitus requiring insulin
14. History of headaches with focal neurological symptoms
15. Uncontrolled thyroid disorder
16. Sickle cell anemia
17. Current or history of clinically significant depression in the last year
18. Known disturbance of lipid metabolism
19. Hepatic adenoma or carcinoma
20. Known or suspected endometrial carcinoma or estrogen-dependent neoplasia
21. Clinically significant history or presence of any gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel diseases, history of cholecystectomy), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting) or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug
22. Difficulty in swallowing study medication
23. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in this study
24. Positive test for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at screening
25. Administration of any investigational drug and/or experimental device within 30 days prior to the screening visit
26. Administration of any biologics within 30 days prior to the screening visit. Note: The Covid-19 vaccine is not included in this prohibition.
27. Clinically significant finding on the ECG suggesting participation in the study could pose a risk to the subject
28. A depot injection or an implant of any drug within 1 month prior to the screening visit
29. Use of oral contraceptives or other sex steroid hormones within 1 month prior to the screening visit. Note: A 1-month drug holiday period is mandatory for potential subjects receiving GnRH agonists and GnRH antagonists.
30. Any clinically significant physical or gynecological abnormality at the screening visit
31. Any clinically significant abnormal laboratory test result at the screening visit
32. Hemoglobin <11.5 g/dL and/or hematocrit <32%
33. Use of over-the-counter products containing any substances which could have the propensity to impact either estradiol or gonadotropin level
34. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing
35. History of seizures, epilepsy, cerebrovascular disorders, central nervous system anomalies or tumors
36. Significant risk factors for decreased bone mineral content and/or bone mass, such as family history (in a first degree relative) of osteoporosis, personal history of chronic use of corticosteroids or anticonvulsants
37. Participation in another drug research within 1 month prior to screening
38. Deemed by the Investigator to have questionable ability to comply with the study protocol, including inadequate adherence to both dosing and use of the AiCure medication adherence monitoring platform during the Run-in Period or during the three Treatment Cycles
39. Current use of any prescription medication known to cause delayed gastric emptying (e.g. glucagon-like peptide-1 receptor agonists)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females, aged 18 to 49 years
Enrollment: 16 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Adequacy of suppression of estradiol (E2) as assessed by the subject incidence of estradiol level below 20 pg/mL | Treatment cycle: Day 29
  The primary PD metric - suppression of E2 level (E2 <20 pg/mL) - will be assessed at each on-treatment evaluation timepoint. E2 below 20 pg/mL at Day 29 is a primary endpoint for a given Treatment Cycle.

SECONDARY OUTCOMES:
Suppression of ovulation (as evidenced by progesterone levels <3 ng/mL) | Treatment cycle: Day 22 and 29
  It will be evaluated with Treatment Cycle Day 22 and Treatment Cycle Day 29 (separately and combined) positioned as most important timepoints for this analyte.
Number of vaginal (menstrual) bleeding days | 28 days of therapy and 14 days post study follow up
  The onset of menstrual period is defined as at least three consecutive bleeding/spotting days during the 14-day postdosing period.
Composite Pelvic Signs and Symptoms (CPSS) scores | Treatment day 29
  CPSS scores (composite and for the individual items) and changes from the pre-dosing baseline will be summarized by treatment received. CPSSS values are derived from the Biberoglu and Behrman scale, with 5 components addressing dysmenorrhea (0-none and 3-severe), dyspareunia (0-none and 3-severe), non-menstrual pelvic pain (0-none and 3-severe), pelvic tenderness (0-none and 3-severe), and pelvic induration (0-none and 3-severe). In composite score (total symptom and sign severity score) 0 being none and 11-15 being very severe.
(Pre-dose leuprolide level) Subject incidence of Leuprolide below detectable level | Treatment Cycle: Days 1, 8, 15, 22 and 29 days
  The summaries will be provided for each PK evaluation timepoint and across the entire treatment cycle
Luteinizing hormone (LH) levels | Treatment days: 1,8, 15, 22 and 29; Post dosing day 14
  Serum concentration measured immediately prior to dosing
Follicle Stimulating Hormone (FSH) levels | Treatment days: 1,8, 15, 22 and 29; Post dosing day 14
  Serum concentration measured immediately prior to dosing

CONTACTS AND LOCATIONS:
Overall Officials: Gary A. Shangold, M.D., Study Chair — Enteris BioPharma Inc.
Locations (4):
- United States (4):
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Complete Healthcare for Women, Columbus, Ohio
  - Tidewater Clinical Research, Norfolk, Virginia
  - Seattle Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No